CLINICAL TRIAL: NCT02952872
Title: Optimizing E-interventions for Alcohol Use: Do Common Factors Apply?
Brief Title: Brief Alcohol E-Interventions Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Emily Grekin, Associate Professor, Wayne State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R21AA023660 (NIH)
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Alcohol Drinking in College
Keywords: Computerized Brief Intervention
MeSH Terms: conditions — Alcohol Drinking in College | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (16):
- Arm 1 (Experimental): Participants will complete a brief tablet-based intervention created to include the following features: no common factors, no human voice, no animated narrator, and no motivational content.
  Interventions: Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use
- Arm 2 (Experimental): Participants will complete a brief tablet-based intervention created to include the following features: no common factors, no human voice, no animated narrator, and motivational content.
  Interventions: Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use
- Arm 3 (Experimental): Participants will complete a brief tablet-based intervention created to include the following features: no common factors, no human voice, the presence of an animated narrator, and no motivational content.
  Interventions: Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use
- Arm 4 (Experimental): Participants will complete a brief tablet-based intervention created to include the following features: no common factors, no human voice, the presence of an animated narrator, and motivational content.
  Interventions: Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use
- Arm 5 (Experimental): Participants will complete a brief tablet-based intervention created to include the following features: no common factors, a human voice guiding the intervention, no animated narrator, and no motivational content.
  Interventions: Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use
- Arm 6 (Experimental): Participants will complete a brief tablet-based intervention created to include the following features: no common factors, a human voice guiding the intervention, no animated narrator, and the presence of motivational content.
  Interventions: Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use
- Arm 7 (Experimental): 7. Participants will complete a brief tablet-based intervention created to include the following features: no common factors, a human voice guiding the intervention, an animated narrator guiding the intervention, and no motivational content.
  Interventions: Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use
- Arm 8 (Experimental): Participants will complete a brief tablet-based intervention created to include the following features: no common factors, a human voice to guide the intervention, an animated narrator to guide the intervention, and the presence of motivational content.
  Interventions: Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use
- Arm 9 (Experimental): Participants will complete a brief tablet-based intervention created to include the following features: common factors, no human voice, no animated narrator, and no motivational content.
  Interventions: Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use
- Arm 10 (Experimental): Participants will complete a brief tablet-based intervention created to include the following features: common factors, no human voice, no animated narrator, and the presence of motivational content.
  Interventions: Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use
- Arm 11 (Experimental): Participants will complete a brief tablet-based intervention created to include the following features: common factors, no human voice, an animated narrator to guide the intervention, and no motivational content.
  Interventions: Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use
- Arm 12 (Experimental): Participants will complete a brief tablet-based intervention created to include the following features: common factors, no human voice, an animated narrator to guide the intervention, and the presence of motivational content.
  Interventions: Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use
- Arm 13 (Experimental): 13. Participants will complete a brief tablet-based intervention created to include the following features: common factors, a human voice to guide the intervention, no animated narrator, and no motivational content.
  Interventions: Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use
- Arm 14 (Experimental): Participants will complete a brief tablet-based intervention created to include the following features: common factors, a human voice to guide the intervention, no animated narrator, and the presence of motivational content.
  Interventions: Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use
- Arm 15 (Experimental): Participants will complete a brief tablet-based intervention created to include the following features: common factors, a human voice to guide the intervention, an animated narrator to guide the intervention, and no motivational content.
  Interventions: Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use
- Arm 16 (Experimental): Participants will complete a brief tablet-based intervention created to include the following features: common factors, a human voice to guide the intervention, an animated narrator to guide the intervention, and the presence of motivational content.
  Interventions: Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use

INTERVENTIONS:
Behavioral: Brief Tablet-based Intervention to Address Heavy Alcohol Use — The intervention will be be tablet-based and take approximately 20 minutes to complete. Content will focus on heavy alcohol use.

SUMMARY:
The project seeks to develop an effective computer-delivered brief intervention to reduce alcohol use using the Multiphase Optimization Strategy (MOST). Sixteen different versions of the intervention will be tested with manipulation of common factors (empathy & positive regard), use of a voice, and use of an animated narrator. Participants will include 352 undergraduate students randomly assigned to one intervention condition; follow-up assessments will take place at one and 3 months. The main outcome will be means drink per day over the past 30 day.

DETAILED DESCRIPTION:
The proposed project seeks to develop a maximally effective computer-delivered brief intervention (CDBI) for reducing heavy alcohol use. To accomplish this, we will use the Multiphase Optimization Strategy (MOST), an efficient method for optimizing intervention content, beginning with factorial designs evaluating main and interaction effects of specific intervention components. Our selection of components will be guided by: (a) Common Factors Theory, which highlights the tremendous contribution of non-specific factors, such as empathy and positive regard, to therapy outcomes, but which is of unknown relevance to CDBIs; and (b) Media Equation Theory, which suggests that people automatically respond to computers in social ways, particularly when those computers replicate human characteristics. To accomplish these goals, we will examine outcomes of computer-delivered brief interventions in which common factors (empathy & positive regard), use of a voice, and use of an animated narrator are systematically manipulated using a factorial design. We will also systematically manipulate the presence vs. absence of motivational content in order to examine possible interactions between common factors and specific motivational techniques. Participants will be 352 undergraduates who are randomly assigned to 1 of 16 intervention conditions. Mean drinks per day over the past 30 days will be measured at 1 and 3-month follow-ups. Secondary analyses will also examine past month heavy drinking days, alcohol-related consequences, and intention to reduce alcohol use. We hypothesize that there will be significant main effects for (1) the factor consistent with Common Factors Theory (empathy and positive regard), (2) the two factors consistent with Media Equation Theory (voice and narrator), and (3) the presence of motivational content. We further hypothesize that mean drinks/day will be lower when (1) the common factors (empathy, positive regard) are combined with a voice and/or narrator or (2) motivational content is combined with common factors and/or a voice/narrator.

ELIGIBILITY:
Inclusion Criteria:

Participants must be students at Wayne State University, aged 18 or older. Additionally, participants must report either (1) consuming 3 (women)/4 (men) drinks per day or 7 (women)/14 (men) drinks per week, (2) getting drunk at least once per week over the past 6 months or (3) binge drinking at least once per week over the past 6 months (i.e. more than 4 (women)/5 (men) drinks in a 2 hr. period).

Exclusion Criteria:

Individuals who are under the age of 18, or who do not meet the study's drinking criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2018-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Grekin, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grekin ER, Beatty JR, McGoron L, Kugler KC, McClure JB, Pop DE, Ondersma SJ. Testing the efficacy of motivational strategies, empathic reflections, and lifelike features in a computerized intervention for alcohol use: A factorial trial. Psychol Addict Behav. 2019 Sep;33(6):511-519. doi: 10.1037/adb0000502. Epub 2019 Aug 22. PMID 31436446

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6 | Arm 7 | Arm 8 | Arm 9 | Arm 10 | Arm 11 | Arm 12 | Arm 13 | Arm 14 | Arm 15 | Arm 16
Started | 22 | 22 | 22 | 22 | 22 | 21 | 22 | 21 | 22 | 22 | 23 | 22 | 22 | 22 | 22 | 23
Completed | 22 | 22 | 22 | 22 | 22 | 21 | 22 | 21 | 22 | 22 | 23 | 22 | 22 | 22 | 22 | 23
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6 | Arm 7 | Arm 8 | Arm 9 | Arm 10 | Arm 11 | Arm 12 | Arm 13 | Arm 14 | Arm 15 | Arm 16 | Total
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22 | 21 | 22 | 21 | 22 | 22 | 23 | 22 | 22 | 22 | 22 | 23 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.68 (3.0) | 24.59 (3.83) | 24.05 (5.92) | 25.91 (4.85) | 24.82 (3.84) | 24.71 (5.36) | 23.82 (2.52) | 27.76 (11.87) | 24.77 (5.55) | 26.18 (8.51) | 23.91 (6.96) | 24 (2.98) | 23.18 (3.54) | 23.95 (2.84) | 23.59 (2.82) | 25.13 (5.82) | 24.62 (5.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 10 | 10 | 13 | 10 | 12 | 6 | 14 | 13 | 12 | 11 | 11 | 10 | 7 | 8 | 173
  Male | 7 | 11 | 12 | 12 | 9 | 11 | 10 | 15 | 8 | 9 | 11 | 11 | 11 | 12 | 15 | 15 | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 3 | 2 | 1 | 0 | 1 | 2 | 0 | 2 | 18
  Not Hispanic or Latino | 20 | 21 | 20 | 22 | 21 | 21 | 21 | 21 | 19 | 20 | 22 | 22 | 21 | 20 | 22 | 21 | 334
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 4 | 4 | 11 | 9 | 3 | 6 | 8 | 6 | 5 | 5 | 7 | 7 | 10 | 5 | 9 | 7 | 106
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 0 | 4 | 1 | 4 | 4 | 3 | 2 | 3 | 2 | 2 | 2 | 0 | 2 | 33
  White | 13 | 15 | 4 | 11 | 12 | 14 | 9 | 11 | 11 | 12 | 10 | 12 | 8 | 12 | 12 | 13 | 179
  More than one race | 3 | 3 | 2 | 1 | 2 | 0 | 1 | 0 | 2 | 3 | 1 | 1 | 1 | 3 | 1 | 1 | 25
  Unknown or Not Reported | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 8
Mean drinks per day [Mean (Standard Deviation); unit: Standard Drinks] | 1.38 (.92) | 1.63 (1.44) | 1.49 (1.57) | 1.94 (2.84) | 1.43 (.92) | 1.71 (1.65) | 1.37 (1.29) | 1.45 (1.06) | 1.36 (1.01) | 1.70 (1.06) | 1.15 (.62) | 1.65 (1.24) | 1.39 (1.36) | 2.20 (1.59) | 1.38 (.97) | 1.50 (1.14) | 1.54 (1.37)

OUTCOME MEASURES:

1. Primary Outcome: Mean Drinks Per Day
Description: Average of reports from past 30 days on the number of standard drinks consumed by participant over the past 30 days.
Time Frame: 1 month and 3 months after baseline
Measure: Mean (Standard Deviation); unit: Drinks per day
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6 | Arm 7 | Arm 8 | Arm 9 | Arm 10 | Arm 11 | Arm 12 | Arm 13 | Arm 14 | Arm 15 | Arm 16
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22 | 21 | 22 | 21 | 22 | 22 | 23 | 22 | 22 | 22 | 22 | 23
Drinks per day
  1 Month Follow-up | .93 (.85) | 1.15 (1.30) | .86 (.97) | 1.38 (1.60) | 1.09 (.88) | 1.17 (1.31) | 1.25 (1.41) | .90 (.78) | 1.70 (2.04) | .94 (.90) | .83 (.45) | 1.19 (1.04) | .96 (1.21) | 1.24 (.86) | 1.02 (1.00) | .88 (.83)
  3 Month Follow-up | .88 (.99) | .79 (.75) | 1.01 (1.17) | 1.02 (1.06) | 1.32 (1.46) | 1.33 (1.81) | 1.09 (.92) | .91 (.87) | 1.87 (2.39) | .59 (.42) | 1.69 (3.45) | 1.02 (1.02) | .75 (.54) | 1.04 (.96) | 1.23 (1.79) | .82 (.75)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4 vs Arm 5 vs Arm 6 vs Arm 7 vs Arm 8 vs Arm 9 vs Arm 10 vs Arm 11 vs Arm 12 vs Arm 13 vs Arm 14 vs Arm 15 vs Arm 16; Test type: Superiority; p < .05, ANOVA; Mixed Design ANOVA

2. Secondary Outcome: Number of Heavy Drinking Days Per Month
Description: Number of days participant reports drinking 4/5 (male/female) alcoholic drinks in a 2-hour period during the past 30 days
Time Frame: 1 month and 3 months after baseline
Measure: Mean (Standard Deviation); unit: Heavy drinking days/month
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6 | Arm 7 | Arm 8 | Arm 9 | Arm 10 | Arm 11 | Arm 12 | Arm 13 | Arm 14 | Arm 15 | Arm 16
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22 | 21 | 22 | 21 | 22 | 22 | 23 | 22 | 22 | 22 | 22 | 23
Heavy drinking days/month
  1 Month Follow-up | 1.86 (2.01) | 2.00 (2.27) | 1.52 (2.00) | 2.05 (2.26) | 2.36 (2.36) | 2.19 (2.29) | 1.64 (1.79) | 1.71 (1.90) | 2.64 (2.63) | 2.32 (2.44) | 2.04 (1.64) | 1.95 (2.17) | 1.59 (1.74) | 2.00 (2.01) | 2.67 (2.54) | 1.78 (2.07)
  3 Month Follow-up | 1.65 (2.35) | 1.76 (2.14) | 1.67 (2.13) | 2.14 (2.40) | 2.45 (2.39) | 2.4 (2.58) | 1.81 (2.34) | 1.65 (2.03) | 2.59 (2.36) | 1.50 (2.09) | 1.96 (1.69) | 2.09 (2.14) | 1.24 (1.67) | 2.18 (2.11) | 2.36 (2.54) | 1.65 (2.13)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4 vs Arm 5 vs Arm 6 vs Arm 7 vs Arm 8 vs Arm 9 vs Arm 10 vs Arm 11 vs Arm 12 vs Arm 13 vs Arm 14 vs Arm 15 vs Arm 16; Test type: Superiority; p < .05, ANOVA

3. Secondary Outcome: Report of Alcohol Related Consequences
Description: Participant self-report on the Brief Young Adult Alcohol Consequences Questionnaire
Time Frame: 1 month and 3 months after baseline
Measure: Mean (Standard Deviation); unit: Alcohol Consequences
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6 | Arm 7 | Arm 8 | Arm 9 | Arm 10 | Arm 11 | Arm 12 | Arm 13 | Arm 14 | Arm 15 | Arm 16
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22 | 21 | 22 | 21 | 22 | 22 | 23 | 22 | 22 | 22 | 22 | 23
Alcohol Consequences
  1 Month Follow-up | 5.24 (5.96) | 3.91 (3.22) | 3.95 (3.80) | 4.41 (4.03) | 5.23 (4.79) | 4.00 (3.18) | 5.23 (4.79) | 3.52 (2.62) | 5.86 (5.22) | 4.91 (4.14) | 3.13 (3.29) | 4.55 (4.32) | 4.00 (4.63) | 4.86 (3.88) | 3.10 (2.64) | 3.96 (2.82)
  3 Month Follow-up | 3.65 (4.72) | 3.67 (3.38) | 3.67 (3.71) | 3.91 (4.60) | 4.36 (4.86) | 3.75 (3.68) | 4.10 (4.42) | 3.00 (4.22) | 4.50 (4.44) | 2.89 (3.07) | 2.78 (2.92) | 4.32 (4.84) | 3.29 (3.85) | 4.18 (3.94) | 2.95 (3.51) | 3.05 (3.11)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4 vs Arm 5 vs Arm 6 vs Arm 7 vs Arm 8 vs Arm 9 vs Arm 10 vs Arm 11 vs Arm 12 vs Arm 13 vs Arm 14 vs Arm 15 vs Arm 16; Test type: Superiority; p < .05, ANOVA

4. Secondary Outcome: Intention to Reduce Alcohol Use
Description: Participants self-report intentions to reduce drinking on the Drinking Intentions Questionnaire. On this questionnaire, participants rate how likely they are to reduce their drinking over the next week, month, and year on a scale ranging from '0 = Not at all likely' to '5 = Extremely likely.' Higher scores mean greater intentions to reduce drinking. In order to obtain more stable estimates and reduce type I error, responses to the week, month and year questions were summed to create a total drinking intentions score which could range from 0 to 15. More specifically, scores on each individual scale item (i.e. intentions to reduce drinking over the week, month and year) could range from 0 to 5. When summed together, these items created the total score (reported here) which could range from 0 to 15.
Time Frame: 1 month and 3 months after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6 | Arm 7 | Arm 8 | Arm 9 | Arm 10 | Arm 11 | Arm 12 | Arm 13 | Arm 14 | Arm 15 | Arm 16
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22 | 21 | 22 | 21 | 22 | 22 | 23 | 22 | 22 | 22 | 22 | 23
score on a scale
  1 Month Follow-up | 6.18 (4.33) | 6.68 (5.01) | 7.48 (5.45) | 8.41 (4.82) | 10.09 (4.31) | 9.29 (4.87) | 7.05 (5.33) | 7.10 (5.06) | 5.09 (3.38) | 8.91 (4.76) | 7.04 (3.90) | 8.00 (4.76) | 7.18 (4.70) | 7.77 (5.14) | 6.52 (4.85) | 6.78 (5.66)
  3 Month Follow-up | 6.50 (4.55) | 6.19 (4.86) | 7.76 (5.06) | 8.36 (5.04) | 10.32 (3.88) | 7.30 (5.35) | 7.81 (5.39) | 6.40 (6.01) | 5.32 (4.13) | 6.39 (5.69) | 6.57 (4.91) | 8.73 (5.01) | 8.76 (4.61) | 8.23 (5.00) | 6.45 (4.89) | 7.29 (6.27)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4 vs Arm 5 vs Arm 6 vs Arm 7 vs Arm 8 vs Arm 9 vs Arm 10 vs Arm 11 vs Arm 12 vs Arm 13 vs Arm 14 vs Arm 15 vs Arm 16; Test type: Superiority; p < .05, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from baseline through the second (3-month post baseline) follow-up.
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6 | Arm 7 | Arm 8 | Arm 9 | Arm 10 | Arm 11 | Arm 12 | Arm 13 | Arm 14 | Arm 15 | Arm 16
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22 | 0/22 | 0/21 | 0/22 | 0/21 | 0/22 | 0/22 | 0/23 | 0/22 | 0/22 | 0/22 | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22 | 0/22 | 0/21 | 0/22 | 0/21 | 0/22 | 0/22 | 0/23 | 0/22 | 0/22 | 0/22 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22 | 0/22 | 0/21 | 0/22 | 0/21 | 0/22 | 0/22 | 0/23 | 0/22 | 0/22 | 0/22 | 0/22 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT02952872/Prot_SAP_000.pdf